CLINICAL TRIAL: NCT02148159
Title: Impact of Mechanism Based Acupuncture Intervention to Improve Weight Loss in GI Cancer Patients With Cachexia
Brief Title: Acupuncture for Unintentional Weight Loss and Anorexia With GI Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB201400340; OCR14647 (Other: University of Florida)
Record Dates: First submitted 2014-05-15; First posted 2014-05-28 (Estimated); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Malignant Neoplasm of Gastrointestinal Tract
Keywords: anorexia; cachexia; cancer; unintentional weigh loss; gastrointestinal tract; adults
MeSH Terms: conditions — Gastrointestinal Neoplasms; Anorexia; Cachexia; Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cachexia Acupuncture-A (Experimental): Acupuncture-A group will receive acupuncture in a pre-determined set of the acupuncture points that are selected based on the potential mechanisms of cachexia. Intervention will be done by a licensed acupuncturist who has over 5 years of experience as an independent clinician and has experience particularly in the management of cancer related symptoms. Acupuncture treatment will consist of 8 sessions over 8 week period.
  Acupuncture needles: Single-use, sterile stainless steel and disposable [acupuncture needles-Peace Classic Needles®, Acu-Market] Other name: Mechanism based acupuncture
  Interventions: Device: Cachexia Acupuncture-A (Peace Classic Needles® )
- General Acupuncture-B (Sham Comparator): General Acupuncture-B group will receive acupuncture in a pre-determined set of the acupuncture points. These points are the real acupuncture points; however, these points are not specific to cachexia management. Participants will receive the acupuncture treatment over 8 weeks (total of 8 sessions) in the same manner as the experimental group; the only difference will be the place(type) and number of points targeted.
  Acupuncture needles: single-use, sterile stainless steel and disposable needles [Peace Classic Needles®, Acu-Market] Other name: General acupuncture
  Interventions: Device: General Acupuncture-B (Peace Classic Needles®)

INTERVENTIONS:
Device: Cachexia Acupuncture-A (Peace Classic Needles® ) — Acupuncture-A group will receive acupuncture in a pre-determined set of the acupuncture points.
  Other Names: Acu-Market; Mechanism based acupuncture
  Arms: Cachexia Acupuncture-A
Device: General Acupuncture-B (Peace Classic Needles®) — Acupuncture-B group will receive acupuncture in a pre-determined set of the acupuncture points.
  Other Names: Acu-Market; General acupuncture
  Arms: General Acupuncture-B

SUMMARY:
Patients with cancer often experience appetite loss and weight loss unintentionally. Rapid weight loss negatively impact on physical functioning, quality of life, and overall survival. Patients will be randomly assigned into two groups. An intervention with acupuncture may slow down or stop the progression of cancer-related anorexia and weight loss.

DETAILED DESCRIPTION:
The purpose of this research study is to investigate if acupuncture helps to improve appetite and slow down unintentional weight loss. The participants will be randomly divided into two groups and receive 8 sessions of acupuncture (two groups will receive different acupuncture points) for 8 weeks. During the study period, participants will be asked various questions about appetite, physical functioning, cancer-related symptoms and quality of life to understand changes related to body weight, as well as blood samples. The research team members will collect data regarding changes in appetite, body weight, body composition, and physical functioning.

ELIGIBILITY:
Inclusion Criteria:

* 21 year or older
* medical diagnosis of gastrointestinal cancer (for example, gastric, biliary, or colorectal)
* experienced weight loss of at least 5% over the last 6 months
* ability to communicate in English
* ability to follow the research protocol

Exclusion Criteria:

* plan to have surgical procedures at the time of recruitment
* receive radiation therapy alone or in addition to chemotherapy during the study period
* undergo surgery during the study or in the months prior to the study
* no plan to have chemotherapy after the surgery
* any comorbidities that may affect the interpretation of study findings
* open burn sites or infected wounds
* esophageal cancer or pancreatic cancer
* life expectancy of less than 6 months as assessed by attending physician

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-10; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Percentage weight change over 8 weeks between two arms | up to 8 weeks
  Weight will be measured each visit (pounds).

SECONDARY OUTCOMES:
Appetite change between two arms | up to 8 weeks
  Three different short survey forms will be used to measure appetite change. Visual analogue scale (0 indicates no appetite and 10 is the best appetite). Simplified Nutritional Appetite Questionnaire score (min-max: 4-20 and the higher the better appetite) Patient Generated Subjective Global Assessment: 0-1, no intervention is needed. 9 or higher score indicates critical intervention.
physical functioning | up to 8 weeks
  survey form (min-max: 0-100, increment by 10%- 100% indicates full functioning).
body composition | up to 8 weeks
  Small, non-invasive device (bioelectrical impedance analysis) like a miniature version of EKG will measure changes in body composition (numeric scale).

OTHER OUTCOMES:
Quality of life between two arms | up to 8 weeks
  Survey format includes the 27 items (5 points scale: 0 means 'not at all' and 4 means 'very much") .
biomarkers | weeks 1, 4 and 8 (three measurements)
  Small amounts of blood will be drawn.
symptom experience | up to 8 weeks
  Survey format: 13 areas related to the symptom experience and patient's concerns will be assessed (4 points scale; 0 means 'not at all' and 3 means 'very much').

CONTACTS AND LOCATIONS:
Overall Officials: Saunjoo Yoon, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Clinical Research Center (CRC), Gainesville, Florida, United States

REFERENCES:
- [Derived] Yoon SL, Grundmann O, Williams JJ, Gordan L, George TJ Jr. Body composition changes differ by gender in stomach, colorectal, and biliary cancer patients with cachexia: Results from a pilot study. Cancer Med. 2018 Aug;7(8):3695-3703. doi: 10.1002/cam4.1665. Epub 2018 Jul 3. PMID 29971962